CLINICAL TRIAL: NCT01235975
Title: Phase IIIb Immunogenicity, Safety and Reactogenicity Study of GSK Biologicals' Meningococcal Vaccine [GSK 134612] When Given as One Dose to Healthy Subjects Aged 56 Years or Older
Brief Title: Immunogenicity and Safety Study of GSK Biologicals' Meningococcal Vaccine Given as One Dose to Healthy Subjects Above 56 Years
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 113807
Record Dates: First submitted 2010-11-04; First posted 2010-11-08 (Estimated); Results first posted 2017-04-28 (Actual); Last update posted 2018-08-20 (Actual); Status verified 2018-07

CONDITIONS: Infections, Meningococcal
Keywords: Neisseria meningitidis; Meningococcal Vaccines; serogroups A,C, W-135 or Y; meningococcal diseases; meningococcal conjugate vaccine; Immunogenicity
MeSH Terms: conditions — Meningococcal Infections

ARMS (2):
- Group A (Experimental)
  Interventions: Biological: Meningococcal vaccine GSK 134612
- Group B (Active Comparator)
  Interventions: Biological: MencevaxACWY TM

INTERVENTIONS:
Biological: Meningococcal vaccine GSK 134612 — Intramuscular injection
  Arms: Group A
Biological: MencevaxACWY TM — Subcutaneous injection
  Arms: Group B

SUMMARY:
This study evaluates the immunogenicity and safety of the meningococcal conjugate vaccine GSK 134612 given as single dose to healthy adults 56 years or older compared to the meningococcal polysaccharide vaccine MencevaxACWYTM.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes can and will comply with the requirements of the protocol
* A male or female 56 years of age or older at the time of the vaccination.
* Written informed consent obtained from the subject.
* Female subjects of non-childbearing potential may be enrolled in the study.
* Non-child-bearing potential is defined as current tubal ligation, hysterectomy, ovariectomy or post-menopause.

Exclusion Criteria:

* Use of any investigational or non-registered product other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Concurrent participation in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or non-investigational product.
* Extended administration of immunosuppressants or other immune-modifying drugs within six months prior to the vaccination. Inhaled and topical steroids are allowed.
* Any contra-indication to intramuscular and /or subcutaneous injection.
* Planned administration/administration of a vaccine not foreseen by the study protocol within 30 days prior to vaccination and ending 30 days after vaccination. (Vaccination with inactivated influenza vaccines, including H1N1, is allowed at any time during the study as per local recommendations).
* Previous vaccination with meningococcal serogroups A, C, W-135 and Y polysaccharide vaccine within 5 years prior to vaccination.
* Previous vaccination at any time with meningococcal serogroups A, C, W-135 and Y polysaccharide conjugate vaccine.
* Previous vaccination with tetanus toxoid containing vaccine within 5 years prior to vaccination.
* History of meningococcal disease due to serogroups A, C, W-135 or Y.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Family history of congenital or hereditary immunodeficiency.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine.
* History of neurological disorders and seizures
* History of Guillain-Barre syndrome.
* Acute (active) clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or pre-existing laboratory screening tests.
* Acute disease and/or fever at the time of enrolment.
* Administration of immunoglobulins and/or any blood products within the 3 months preceding the first dose of study vaccine/product or planned administration during the study period.
* Pregnant or lactating female.
* Current chronic alcohol consumption and/or drug abuse.

Min Age: 56 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2010-11-30 (Actual); Primary Completion 2011-07-29 (Actual); Study Completion 2011-08-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Dbaibo G, El-Ayoubi N, Ghanem S, Hajar F, Bianco V, Miller JM, Mesaros N. Immunogenicity and safety of a quadrivalent meningococcal serogroups A, C, W-135 and Y tetanus toxoid conjugate vaccine (MenACWY-TT) administered to adults aged 56 Years and older: results of an open-label, randomized, controlled trial. Drugs Aging. 2013 May;30(5):309-19. doi: 10.1007/s40266-013-0065-0. PMID 23494214
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 113807 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113807 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113807 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113807 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113807 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113807 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of the total number of subjects originally enrolled, only 369 subjects were eventually found to be eligible to be included in the Total Vaccinated Cohort.
Groups:
- Nimenrix Group: Healthy male or female subjects aged 56 years or older received a single dose of Nimenrix conjugate vaccine, administered intramuscularly into the deltoid region of the non-dominant arm, at Day 0.
- Mencevax Group: Healthy male or female subjects aged 56 years or older received a single dose of Mencevax vaccine, administered by subcutaneous injection in the upper region of the non-dominant arm, at Day 0.
Period: Overall Study
Arm/Group | Nimenrix Group | Mencevax Group
Started | 274 | 95
Completed | 257 | 88
Not Completed | 17 | 7
Not completed — Serious Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 8 | 2
Not completed — Migrated/moved from study area | 2 | 1
Not completed — Lost to Follow-up | 7 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nimenrix Group | Mencevax Group | Total
Number analyzed (Participants) | 274 | 95 | 369
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.1 (7.22) | 64.3 (7.39) | 64.15 (7.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 182 | 70 | 252
  Male | 92 | 25 | 117
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White - Arabic / North African Heritage | 274 | 95 | 369

OUTCOME MEASURES:

1. Primary Outcome: Vaccine Response to Meningococcal Antigens (MenA, MenC, MenW-135 and MenY)
Description: Vaccine response for serum bactericidal assay using rabbit complement (rSBA) antibodies against Neisseria meningitides serogroups A, C , W-135, Y (rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY) was defined as: for initially seronegative subjects [rSBA titer below (<) 1:8], post-vaccination rSBA titer greater than or equal to (≥) 1: 32; for initially seropositive subjects with rSBA titer between 1:8 and 1:128, at least four-fold increase in rSBA titer from pre to post vaccination; and for initially seropositive subjects with rSBA titer ≥1:128, at least two-fold increase in rSBA titer from pre to post vaccination.
Time Frame: One month after vaccination (Month 1)
Population: The primary analysis was performed on the According-to-protocol (ATP) cohort for immunogenicity, which included all evaluable subjects who met all eligibility criteria, who complied with the protocol requirements and for whom immunogenicity measures were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Mencevax Group
Number analyzed (Participants) | 188 | 66
Participants
  rSBA-MenA: number analyzed (Participants) | 175 | 60
  rSBA-MenA | 134 | 55
  rSBA-MenC | 151 | 56
  rSBA-MenW-135: number analyzed (Participants) | 187 | 62
  rSBA-MenW-135 | 145 | 54
  rSBA-MenY: number analyzed (Participants) | 188 | 64
  rSBA-MenY | 154 | 57

2. Secondary Outcome: Number of Subjects With rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY Antibody Titers ≥ the Cut-off Value
Description: The cut-off value for the rSBA titers was greater than or equal to (≥) 1:8.
Time Frame: At Day 0 and Month 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Mencevax Group
Number analyzed (Participants) | 193 | 66
Participants
  rSBA-MenA, Day 0: number analyzed (Participants) | 181 | 61
  rSBA-MenA, Day 0 | 136 | 43
  rSBA-MenA, Month 1: number analyzed (Participants) | 186 | 65
  rSBA-MenA, Month 1 | 185 | 65
  rSBA-MenC, Day 0: number analyzed (Participants) | 190 | 66
  rSBA-MenC, Day 0 | 135 | 44
  rSBA-MenC, Month 1: number analyzed (Participants) | 192 | 66
  rSBA-MenC, Month 1 | 192 | 65
  rSBA-MenW-135, Day 0: number analyzed (Participants) | 188 | 62
  rSBA-MenW-135, Day 0 | 135 | 40
  rSBA-MenW-135, Month 1 | 188 | 63
  rSBA-MenY, Day 0: number analyzed (Participants) | 189 | 64
  rSBA-MenY, Day 0 | 148 | 55
  rSBA-MenY, Month 1 | 193 | 66

3. Secondary Outcome: Number of Subjects With rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY Antibody Titers ≥ the Cut-off Value
Description: The cut-off value for the rSBA titers was greater than or equal to (≥) 1:128.
Time Frame: At Day 0 and Month 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Mencevax Group
Number analyzed (Participants) | 193 | 66
Participants
  rSBA-MenA, Day 0: number analyzed (Participants) | 181 | 61
  rSBA-MenA, Day 0 | 104 | 37
  rSBA-MenA, Month 1: number analyzed (Participants) | 186 | 65
  rSBA-MenA, Month 1 | 177 | 63
  rSBA-MenC, Day 0: number analyzed (Participants) | 190 | 66
  rSBA-MenC, Day 0 | 86 | 29
  rSBA-MenC, Month 1: number analyzed (Participants) | 192 | 66
  rSBA-MenC, Month 1 | 179 | 62
  rSBA-MenW-135, Day 0: number analyzed (Participants) | 188 | 62
  rSBA-MenW-135, Day 0 | 98 | 30
  rSBA-MenW-135, Month 1 | 183 | 62
  rSBA-MenY, PRE Day 0: number analyzed (Participants) | 189 | 64
  rSBA-MenY, PRE Day 0 | 118 | 46
  rSBA-MenY, Month 1 | 187 | 65

4. Secondary Outcome: rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY Antibody Titers
Description: Antibody titers were presented as geometric mean titers (GMTs).
Time Frame: At Day 0 and Month 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Nimenrix Group | Mencevax Group
Number analyzed (Participants) | 193 | 66
Titers
  rSBA-MenA, Day 0: number analyzed (Participants) | 181 | 61
  rSBA-MenA, Day 0 | 108.3 [77.9 to 150.5] | 102.1 [55.2 to 188.7]
  rSBA-MenA, Month 1: number analyzed (Participants) | 186 | 65
  rSBA-MenA, Month 1 | 1442.3 [1174.4 to 1771.3] | 2840.1 [2062.3 to 3911.1]
  rSBA-MenC, Day 0: number analyzed (Participants) | 190 | 66
  rSBA-MenC, Day 0 | 71.5 [51.1 to 100.1] | 73.8 [38.0 to 143.6]
  rSBA-MenC, Month 1: number analyzed (Participants) | 192 | 66
  rSBA-MenC, Month 1 | 2498.6 [1887.0 to 3308.2] | 4815.1 [2827.0 to 8201.2]
  rSBA-MenW-135, Day 0: number analyzed (Participants) | 188 | 62
  rSBA-MenW-135, Day 0 | 84.7 [61.1 to 117.3] | 68.5 [37.4 to 125.3]
  rSBA-MenW-135, Month 1 | 1454.0 [1130.5 to 1870.1] | 1838.4 [1134.6 to 2978.9]
  rSBA-MenY, Day 0: number analyzed (Participants) | 189 | 64
  rSBA-MenY, Day 0 | 137.6 [100.7 to 187.9] | 217.4 [131.7 to 358.9]
  rSBA-MenY, Month 1 | 2547.0 [2059.6 to 3149.8] | 3931.6 [2726.1 to 5670.2]

5. Secondary Outcome: Number of Subjects With Anti-polysaccharide Meningococcal Serogroup A (Anti-PSA), Serogroup C (Anti-PSC), Serogroup W-135 (Anti-PSW-135) and Serogroup Y (Anti-PSY) Antibody Concentrations ≥ the Cut-off Value
Description: The cut-off value for the anti-polysaccharide concentrations was greater than or equal to (≥) 0.3 micrograms per milliliter (μg/mL).
Time Frame: At Day 0 and Month 1
Population: The primary analysis was performed on a subset of of the 2 treatment groups and 2 age strata of the According-to-protocol (ATP) cohort for immunogenicity, 50% of subjects were tested for anti-PSA and anti-PSC and the other 50% of subjects were tested for anti-PSW-135 and anti-PSY.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Mencevax Group
Number analyzed (Participants) | 75 | 27
Participants
  anti-PSA, Day 0: number analyzed (Participants) | 71 | 24
  anti-PSA, Day 0 | 66 | 23
  anti-PSA, Month 1: number analyzed (Participants) | 73 | 25
  anti-PSA, Month 1 | 72 | 25
  anti-PSC, Day 0: number analyzed (Participants) | 75 | 26
  anti-PSC, Day 0 | 51 | 23
  anti-PSC, Month 1: number analyzed (Participants) | 75 | 26
  anti-PSC, Month 1 | 73 | 26
  anti-PSW-135, Day 0: number analyzed (Participants) | 67 | 27
  anti-PSW-135, Day 0 | 46 | 16
  anti-PSW-135, Month 1: number analyzed (Participants) | 57 | 24
  anti-PSW-135, Month 1 | 54 | 24
  anti-PSY, Day 0: number analyzed (Participants) | 64 | 25
  anti-PSY, Day 0 | 43 | 18
  anti-PSY, Month 1: number analyzed (Participants) | 61 | 25
  anti-PSY, Month 1 | 60 | 25

6. Secondary Outcome: Number of Subjects With Anti-PSA, Anti-PSC, Anti-PSW-135 and Anti-PSY Antibody Concentrations ≥ the Cut-off Value
Description: The cut-off value for the anti-polysaccharide concentrations was greater than or equal to (≥) 2.0 micrograms per milliliter (μg/mL).
Time Frame: At Day 0 and Month 1
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Mencevax Group
Number analyzed (Participants) | 75 | 27
Participants
  anti-PSA, Day 0: number analyzed (Participants) | 71 | 24
  anti-PSA, Day 0 | 43 | 14
  anti-PSA, Month 1: number analyzed (Participants) | 73 | 25
  anti-PSA, Month 1 | 66 | 23
  anti-PSC, Day 0: number analyzed (Participants) | 75 | 26
  anti-PSC, Day 0 | 24 | 10
  anti-PSC, Month 1: number analyzed (Participants) | 75 | 26
  anti-PSC, Month 1 | 63 | 25
  anti-PSW-135, Day 0: number analyzed (Participants) | 67 | 27
  anti-PSW-135, Day 0 | 22 | 4
  anti-PSW-135, Month 1: number analyzed (Participants) | 57 | 24
  anti-PSW-135, Month 1 | 43 | 22
  anti-PSY, Day 0: number analyzed (Participants) | 64 | 25
  anti-PSY, Day 0 | 9 | 5
  anti-PSY, Month 1: number analyzed (Participants) | 61 | 25
  anti-PSY, Month 1 | 51 | 23

7. Secondary Outcome: Anti-PSA, Anti-PSC, Anti-PSW-135 and Anti-PSY Antibody Concentrations
Description: Antibody concentrations were presented as geometric mean concentrations (GMCs), expressed in micrograms per milliliter (μg/mL).
Time Frame: At Day 0 and Month 1
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Nimenrix Group | Mencevax Group
Number analyzed (Participants) | 75 | 27
μg/mL
  anti-PSA, Day 0: number analyzed (Participants) | 71 | 24
  anti-PSA, Day 0 | 3.62 [2.42 to 5.41] | 5.35 [2.36 to 12.11]
  anti-PSA, Month 1: number analyzed (Participants) | 73 | 25
  anti-PSA, Month 1 | 22.92 [15.02 to 34.97] | 57.67 [26.37 to 126.10]
  anti-PSC, Day 0: number analyzed (Participants) | 75 | 26
  anti-PSC, Day 0 | 0.96 [0.66 to 1.40] | 1.46 [0.81 to 2.66]
  anti-PSC, Month 1: number analyzed (Participants) | 75 | 26
  anti-PSC, Month 1 | 8.97 [6.21 to 12.97] | 22.50 [13.80 to 36.66]
  anti-PSW-135, Day 0: number analyzed (Participants) | 67 | 27
  anti-PSW-135, Day 0 | 1.01 [0.65 to 1.58] | 0.77 [0.34 to 1.73]
  anti-PSW-135, Month 1: number analyzed (Participants) | 57 | 24
  anti-PSW-135, Month 1 | 9.01 [5.39 to 15.08] | 24.02 [11.18 to 51.61]
  anti-PSY, Day 0: number analyzed (Participants) | 64 | 25
  anti-PSY, Day 0 | 0.56 [0.41 to 0.77] | 0.88 [0.42 to 1.85]
  anti-PSY, Month 1: number analyzed (Participants) | 61 | 25
  anti-PSY, Month 1 | 11.47 [7.32 to 17.97] | 19.64 [9.53 to 40.50]

8. Secondary Outcome: Number of Subjects With Anti-tetanus Toxoid (Anti-TT) Antibody Concentrations ≥ the Cut-off Value
Description: The cut-off value for the anti-TT concentrations was greater than or equal to (≥) 0.1 international units per milliliter (IU/mL).
Time Frame: At Day 0 and Month 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Mencevax Group
Number analyzed (Participants) | 192 | 66
Participants
  Anti-TT, Day 0 | 12 | 6
  Anti-TT, Month 1 | 54 | 6

9. Secondary Outcome: Anti-tetanus Toxoid (Anti-TT) Antibody Concentrations
Description: Antibody concentrations were presented as geometric mean concentrations (GMCs), expressed in international units per milliliter (IU/mL).
Time Frame: At Day 0 and Month 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Nimenrix Group | Mencevax Group
Number analyzed (Participants) | 192 | 66
IU/mL
  anti-TT, Day 0 | 0.058 [0.053 to 0.063] | 0.060 [0.051 to 0.070]
  anti-TT, Month 1 | 0.137 [0.104 to 0.180] | 0.060 [0.051 to 0.071]

10. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = significant pain at rest or pain that prevented normal every day activities. Grade 3 redness/swelling = redness/swelling spreading beyond 50 millimeters (mm) of injection site.
Time Frame: Within 4 days (Day 0 to 3) post-vaccination
Population: The primary analysis was performed on the Total Vaccinated Cohort (TVC), which included all subjects with vaccine administration documented, who had filled in their symptom sheets.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Mencevax Group
Number analyzed (Participants) | 265 | 89
Participants
  Any Pain | 6 | 0
  Grade 3 Pain | 0 | 0
  Any Redness | 3 | 0
  Grade 3 Redness | 0 | 0
  Any Swelling | 3 | 0
  Grade 3 Swelling | 0 | 0

11. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were fatigue,gastrointestinal symptoms, headache and temperature [defined as orally temperature equal to or above (≥) 37.5 degrees Celsius (°C)]. Any = occurrence of any general symptom regardless of intensity grade or relationship to vaccination. Grade 3 symptom = symptom that prevented normal activity. Grade 3 temperature = temperature above (>) 39.5 °C. Related = symptom assessed by the investigator as causally related to the study vaccination.
Time Frame: Within 4 days (Day 0 to 3) post-vaccination
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Mencevax Group
Number analyzed (Participants) | 265 | 89
Participants
  Any Fatigue | 5 | 0
  Grade 3 Fatigue | 0 | 0
  Related Fatigue | 3 | 0
  Any Gastrointestinal symptoms | 0 | 0
  Grade 3 Gastrointestinal symptoms | 0 | 0
  Related Gastrointestinal symptoms | 0 | 0
  Any Headache | 8 | 2
  Grade 3 Headache | 0 | 0
  Related Headache | 6 | 1
  Any Temperature (Orally) | 6 | 1
  Grade 3 Temperature (Orally) | 0 | 0
  Related Temperature (Orally) | 3 | 0

12. Secondary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: Within 31 days (Day 0 to 30) after vaccination
Population: The primary analysis was performed on the Total Vaccinated cohort (TVC), which cohort included all subjects with vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Mencevax Group
Number analyzed (Participants) | 274 | 95
Participants | 1 | 2

13. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: Within 31 days (Day 0 to 30) after vaccination
Population: The primary analysis was performed on the Total Vaccinated Cohort (TVC), which included all subjects with vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Mencevax Group
Number analyzed (Participants) | 274 | 95
Participants | 0 | 1

14. Secondary Outcome: Number of Subjects With New Onset Chronic Illnesses (NOCI)
Description: NOCIs include autoimmune disorders, asthma, type I diabetes, allergies.
Time Frame: Within 31 days (Day 0 to 30) after vaccination
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group | Mencevax Group
Number analyzed (Participants) | 274 | 95
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Solicited local/general symptoms during the 4-day post-vaccination period (Days 0-3), Unsolicited AEs during the 31-day post-vaccination (Days 0-30), SAEs during the entire study period (from Day 0 up to Month 1).
Description: All frequent adverse events reported were below the 5% frequency threshold.
Arm/Group | Nimenrix Group | Mencevax Group
All-Cause Mortality (participants affected / at risk) | 0/274 | 0/95
Serious Adverse Events (participants affected / at risk) | 0/274 | 1/95
Other Adverse Events (participants affected / at risk) | 0/274 | 0/95
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nimenrix Group (N=274) | Mencevax Group (N=95)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.